CLINICAL TRIAL: NCT05424120
Title: Thoracentesis Quality Improvement (QI) Study
Brief Title: Thoracentesis QI Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PACCS-2021-30297
Record Dates: First submitted 2022-04-25; First posted 2022-06-21 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Pleural Effusion
Keywords: pleural effusion; thoracentesis; wall suction; manual aspiration; vacuum bottle drainage
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled, non-blinded, single-center, quality improvement study to determine which method of standard of care thoracentesis (wall suctioning, manual aspiration, or vacuum drainage) has the shortest procedural time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Manual aspiration (Active Comparator): pleural fluid is drained using a standard thoracentesis kit and via a syringe and three-way stopcock
  Interventions: Procedure: Manual aspiration
- Wall suction (Active Comparator): pleural fluid is drained using a standard thoracentesis kit and by attaching tubing to wall suctioning set at -50 mmHg continuously
  Interventions: Procedure: Wall suction
- Vacuum bottle drainage (Active Comparator): pleural fluid is drained using a standard thoracentesis kit and tubing that attaches to a glass vacuum container
  Interventions: Procedure: Vacuum bottle drainage

INTERVENTIONS:
Procedure: Manual aspiration — One option from standard of care
  Arms: Manual aspiration
Procedure: Wall suction — One option from standard of care
  Arms: Wall suction
Procedure: Vacuum bottle drainage — One option from standard of care
  Arms: Vacuum bottle drainage

SUMMARY:
Researchers will compare 3 standard of care methods of pleural fluid drainage during therapeutic thoracentesis. Patients are randomized to manual aspiration, vacuum bottle drainage or wall suction methods. Primary outcome is procedural time with secondary outcomes of pain and dyspnea scores.

ELIGIBILITY:
Inclusion Criteria:

* Age >18
* Evidence of pleural effusion on imaging
* Clinical indication for thoracentesis

Exclusion Criteria:

* Age <18
* Standard contraindication for thoracentesis procedure
* Patients on positive pressure ventilation
* Patients who have opted out of research in EPIC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Procedural time to 500mL | Through study completion, an average of 24 hours
  Time to pleural fluid drainage from initiation of therapeutic drainage to 500mL
Procedural time to 750mL | Through study completion, an average of 24 hours
  Time to pleural fluid drainage from initiation of therapeutic drainage to 750mL
Procedural time to 1L | Through study completion, an average of 24 hours
  Time to pleural fluid drainage from initiation of therapeutic drainage to 1L
Pain and dyspnea scores- Baseline | Immediately prior to starting the thoracentesis
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)
Pain and dyspnea scores- Cath | Through study completion, an average of 24 hours
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)
Pain and dyspnea scores- Post-fluid | Through study completion, an average of 24 hours
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)
Pain and dyspnea scores- Post-cath | Immediately after removing the thoracentesis catheter
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)
Pain and dyspnea scores- 5m post | 5 minutes post-procedure
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)
Pain and dyspnea scores- 24h post | 24 hours post-procedure
  Patients will be asked to indicate their pain and dyspnea level verbally using the Modified Borg Scale for Dyspnea and Numerical Ratings Scale (0-10, with 10 being highest level of pain)

CONTACTS AND LOCATIONS:
Overall Officials: Roy Cho, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States